CLINICAL TRIAL: NCT04763577
Title: Prognostic Value of the Bradykinin-degradating Enzymes Activities on the Relapse Risk of Angiotensin-Converting Enzyme Inhibitors-associated Angioedema
Brief Title: Bradykinin-degradating Enzymes Activities in Angiotensin-Converting Enzyme Inhibitors-associated Angioedema
Acronym: KIN-ACE
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Collaborators: University Hospital, Paris (Other); University Hospital, Rouen (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC19.025; 2020-A00775-34 (Other: ID RCB)
Record Dates: First submitted 2021-02-16; First posted 2021-02-21 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Angio-Oedema Caused by Angiotensin-Converting-Enzyme Inhibitor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Citrate plasma sample serum sample EDTA sample
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Assay of Bradykinin-degradating enzymes. — Aminopeptidase P activity assay; Dipeptidyl peptidase IV activity assay; Angiotensin Converting Enzyme activity assay; MME gene polymorphisme exploration.

SUMMARY:
Angiotensin-Converting-Enzyme-inhibitors-dependent angioedema (ACEi-AE) is the most frequent form of bradykinin-mediated AE, with an estimated prevalence of 0.1% to 0.7%.

These AE can be explained by the accumulation of bradykinin (BK), a peptide responsible for increase of vascular permeability: ACE inhibitors block ACE, the main inactivation pathway of the BK, thus extending its half-life.

In spite of the the stopping of the drug, systematically performed in the case of ACEi-AE, up to 50% of patients relapsed within 6 months, with maximum risk in the first month after stopping. In addition, the discontinuation of these drugs represents a loss of chance for some patients, without clearly established mastocytic (or histaminic) or bradykinic etiology.

At present there is no method to predict the risk of crisis recurrence in patients who have developed AE-IEC.

The investigators hypothesize that the risk of relapse is associated with a decrease in the activity of BK degradation enzymes (including aminopeptidase P (APP), dipeptidyl peptidase-4 (DPP4), and ECA) that persists at the cessation of IEC.

ELIGIBILITY:
Inclusion Criteria:

* Men and women at least 18 years old
* Presenting AE secondary to treatment with Angiotensin Conversion Enzyme Inhibitors for less than 15 days, or an isolated AE (without superficial hives), which lasts at least 15 hours, and whose diagnosis is validated by the expert committee,
* Having signed informed and written consent
* And being affiliated with social security

Exclusion Criteria:

* Patient who had one or more AEs prior to IEC
* Hereditary or acquired deficiency of C1 inhibitor
* Subject with known mutation of the F12 or PLG gene Subject in times of exclusion from another research involving the human person type 1 or 2 Persons referred to in sections L1121-5 to L1121-8 of the public health code (pregnant woman, breastfeeding mother, person deprived of liberty, person subject to legal protection) subject that cannot be contacted in an emergency situation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Angioedema secondary to Angiotensin Converting Enzyme Inhibitors
Sampling Method: Non-Probability Sample
Enrollment: 243 (Estimated)
Dates: Start 2021-10-27 (Actual); Primary Completion 2025-10-26 (Estimated); Study Completion 2025-10-26 (Estimated)

PRIMARY OUTCOMES:
Prognostic Value of Bradykinin degradating enzymes | Association between the activity of kinin-degrading enzymes (ECA, APP, DPP4) measured by enzyme methods, expressed in tertiles, and relapse at 6 months.
  The primary outcome is to determine the dynamic prognostic value of each of the kinin catabolism enzyme activities, as biomarkers of the risk of relapse at 6 months in patients with BK-AE associated with ACEi.

CONTACTS AND LOCATIONS:
Overall Officials: Federica DEFENDI, Principal Investigator — University Hospital, Grenoble
Locations (4):
- France (4):
  - Chu Grenoble Alpes, Grenoble
  - CHRU de Lille _Hôpital Claude-Huriez, Lille
  - AP-HP _St Antoine, Paris
  - CHU de Rouen, Rouen